CLINICAL TRIAL: NCT06870097
Title: An 8 Week, Stratified Randomiz Ation , Double Blind , Crossover , Placebo Controlled Trial for the Evaluation of the the Effects of A2 Milk on Gut Beneficial Bacteria Growth, Antioxidant Activity, Digestion, and Inflammation Improvement
Brief Title: A Study on the Effects of A2 Milk on Gut Beneficial Bacteria Growth and Digestion Improvement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: B-2412-943-002
Record Dates: First submitted 2025-02-28; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Digestive Discomfort

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A2 Milk (Active Comparator): A2 milk, 275 mL, twice daily after meal (550 mL/day)
  Interventions: Other: A2 Milk
- A1/A2 milk (Placebo Comparator): A1/A2 milk, 275 mL, twice daily after meal (550 mL/day)
  Interventions: Other: A1/A2 Milk

INTERVENTIONS:
Other: A2 Milk — Cow's milk that contains only A2 β-Casein
  Arms: A2 Milk
Other: A1/A2 Milk — Cow's milk that contains both A1 β-Casein and A2 β-Casein
  Arms: A1/A2 milk

SUMMARY:
The aim of this study is to evaluate the effects of A2 milk on gut beneficial bacteria growth, antioxidant activity , digestion, and inflammation improvement

DETAILED DESCRIPTION:
Milk has a high calcium content, and calcium in milk is easily digested and absorbed and has an excellent utilization rate in the body. Milk is rich in lactose, Vitamin D, and peptides that facilitate calcium absorption, and it also contains essential amino acids and bioactive substances that are beneficial to health. Regularly drinking milk has been proven to improve insulin sensitivity, blood pressure, and serum lipid concentrations. Furthermore, milk is reported to be an effective food for nutritional supplementation and improvement in the diet of Koreans, as it contains a well balanced source of essential amino acids that can be lacking in a rice centric diet, along with quality animal protein, calcium, vitamin B2, and other nutrients. However, this increase in dairy consumption can be associated with an increased risk for certain disorders, including digestive disorders.

The actual prevalence of lactose intolerance is unclear in Korea, and reports have ranged from 39.1% to 84.1%. In 2010, it was reported that in most individuals who believed they had lactose intolerance, no evidence of problems with lactose absorption could be found, and thus, gastrointestinal symptoms were unlikely to be associated with lactose. Alternatively, A1 β-Casein and β-Casomorphin-7 (BCM-7) has emerged as a major area for research in relation to digestive discomfort following milk consumption.

Milk is composed of 80% Casein protein and 20% whey. Among Casein proteins, β-Casein can be divided into the A1 type comprised of A1, B, C, F, and G, and the A2 type with A2, A3, D, E, H, I, and J variants. A1 and A2 type β-Casein proteins differ in their 67th amino acid, with A1 containing Histidine and B2 with Proline.

The other remaining variants are only found in low levels or not found in European cattle. Furthermore, BCM-7, which is produced when enzymatic cleavage at the histidine position occurs in A1 β-Casein, has been associated with digestive discomfort. Additionally, milk containing A1 β-Casein has been linked to type 1 diabetes and heart disease. Nevertheless, the majority of dairy cattle in dairy industries continue to produce milk containing A1 β-Casein.

Animal tests have shown that milk with A1 β-Casein takes longer to transit through the digestive tract compared to A2 β-Casein containing milk. In addition, a clinical trial reported that the Bristol stool scores in participants who consumed A1 β-Casein milk were higher than those in A2 β-Casein milk. Another clinical trial announced that A2 β-Casein milk alleviated gastrointestinal symptoms of milk hypersensitivity. In addition, there are reports that blood GSH levels, intestinal short chain fatty acids (Acetic acid, butanoic acid), and intestinal beneficial bacteria (Bifidobacterium genus) content are increased.

Therefore, this study aims to evaluate the effects of A2 milk on gut beneficial bacteria growth, antioxidant activity , digestion, and inflammation improvement compared to a control (A1/A2 milk) in individuals who experience discomfort after consuming milk.

ELIGIBILITY:
Inclusion Criteria:

* Between 19 to 65 years of age
* Participants who are experiencing digestive symptoms abdominal bloating, abdominal pain, borborygmus, fecal urgency, flatulence, diarrhea, nausea) following milk consumption on Visit 1 with a total score on the digestive discomfort symptom survey being 7 point or more for the following 5 items: abdominal pain, borborygmus , flatulence, diarrhea, nausea. (Individuals who have indicated scored 7 or more on any one item in the symptom will be excluded)
* Those who have agreed to participate and given written consent through the Informed Consent Form prior to the study

Exclusion Criteria:

* Currently undergoing treatment for severe cardiovascular, immune, respiratory, gastrointestinal/hepatic and biliary, renal an durinary, neurological, musculoskeletal, mental, infectious, metabolic diseases, and malignancies
* Diagnosed with or has a history of gastrointestinal diseases (irritable bowel syndrome, colitis, ulcerative colitis, abdominal diseases etc.), or has undergone gastrointestinal surgery
* History of bowel obstruction
* Hospitalized within the last 3 months of Visit 1
* Has taken the following drugs or foods within 3 months of visit 1

  ① Drugs that affect body weight {obesity drugs (appetite suppressants, fat absorption inhibitors, Glucagon-like peptide-1 (GLP-1) recept or agonists etc.) etc.), diabetes drugs, etc.}

  ② Psychiatric drugs such as antidepressants and antipsychotics

  ③ Diuretics

  ④ Systemic steroid preparations and hormonal preparations (including oral contraceptives and thyroid hormone preparations
* Has taken immunosuppressive drugs or anti inflammatory drugs within the last month (30 days) of Visit 1
* Administered systemic antibiotics, systemic antibacterial agents, colonics, bowel cleansers, probiotics, prebiotics, antioxidant related health functional foods (Coenzyme Q10, red ginseng, etc.), and glutathione containing products within 2 weeks of visit 1 (however, vitamin preparations can be used together if taken without changing dosage or medication for more than 3 months
* Has taken prokinetics (Serotonin type 4 (5-HT4) Agonist, D2 Antagonists, Cholinergic Agonists etc.), laxatives {fiber supplements (Psyllium, Methylce llulose etc.), stool softeners, osmotic laxatives (Sorbitol, Lactulose etc.), stimulant laxatives (Bisacodyl , Anthraquinone etc.)} within 1 week of visit 1
* History of alcohol abuse or who chronically consume alcohol*

  * Drinking alcohol equivalent to an average of 40 g or more per day (280 g/week) for men and more than 20 g of alcohol per day (140 g/we ek) for women.
* Pregnant, breastfeeding, or planning to become pregnant during the study period
* Participated in another interventional clinical trial (including human trials) within the last 3 months of Visit 1, or planning to participate in another interventional clinical trial (including human trials) after the start of this study
* Allergic to dairy products (bloody stool, muscle/joint pain, headache, dizziness, coma, short term memory impairment, oral ulcer, cardiac arrhythmia, sore throat, increased frequency of urination, acne, depression)
* Individuals deemed inappropriate for the study by the investigator

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale (GSRS) Total Score | Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  Evaluated through the Gastrointestinal Symptom Rating Scale (GSRS) which uses a 7 point Likert type scale from 1 (no symptoms or normal) to 7(severe symptoms) to rate 15 symptom items including both upper and lower abdominal symptoms. Participants will be given the GSRS to complete.

SECONDARY OUTCOMES:
Digestive Discomfort Symptom Survey | Surveys given on Screening(week -2), Visit 3(week 2) to recorded once a day; Retrieved on Visit 2(week 0), Visit 4(week 4) to recorded twice a day within 30 minutes to 3 hours after consuming the test food;
  Participants rate 7 items (abdominal bloating, abdominal pain, borborygmus , fecal urgency, flatulence, diarrhea, nausea) on a numeral rating scale of 0 (Never) to 10 (Very Severe).
Visual analogue scale Irritable Bowel Syndrome (VAS-IBS) | Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  The scale of symptoms felt by 7 items {abdominal symptoms (abdominal pain, diarrhea, constipation, abdominal bloating or flatulence , nausea or vomiting) and health and daily items} is displayed on a 100 mm straight line from 0 mm (very good) to 100 mm (very severe).
Blood Marker : Glutathione (GSH) | Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  Serum levels of GSH measured in ug/mL
Blood Marker : 8-Oxo-2'-deoxyguanosine (8-OxodG) | Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  Serum levels of 8-OxodG measured in ng/mL
Blood Marker : 5-hydroxymethyl-deoxyuridine (5-OHmdU) | Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  Serum levels of 5-OHmdU measured in ng/mL
Blood Marker : High Sensitive C-reactive protein (hs-CRP) | Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  Serum levels of hs-CRP measured in mg/dL
Blood marker : Interleukin-4 (IL-4) | Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  Serum levels of IL-4 measured in pg/mL.
Blood marker : Interleukin-6 (IL-6) | Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  Serum levels of IL-6 measured in pg/mL
Blood Marker : Tumor necrosis factor-α (TNF-α) | Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  Serum levels of TNF-α measured in pg/mL.
Blood Marker : Dipeptidyl Peptidase-4 (DPP-IV) | Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  Serum levels of DPP-IV measured in ng/mL.
Blood Marker : β-casomorphin-7 (BCM-7) | Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  Serum levels of BCM-7 measured in ug/mL.
Blood Marker : β casomorphin-10 (BCM-10) | Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  Serum levels of BCM-10 measured in ug/mL.
Stool marker : Short chain Fatty Acid (SCFA) | Stool collection kit provided on Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4); Retrieved on Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  SCFA in stool measured in mg/g.
Stool marker : Calprotectin | Stool collection kit provided on Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4); Retrieved on Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  Calprotectin in stool measured in mg/kg.
Stool marker : Microbiome | Stool collection kit provided on Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4); Retrieved on Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  Gut microbiome composition (abundance, %) will be measured in stool via 16S ribosomal ribonucleic acid (rRNA)
Bowel Frequency and Form | Journal provided on Screening (week -2), Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4) to record daily; Retrieved on Visit 2 (week 0), Visit 3 (week 2), Visit 4 (week 4), Visit 5 (week 6)
  Participants record daily bowel frequency and form. The Bristol Stool Scale will be used to measure stool consistency with type 1 (Separate hard lumps, like nuts hard to pass), type 2 (Sausage shaped but lumpy), type 3 (Like a sausage but with cracks on its surface), type 4 (Like a sausage or snake, smooth and soft), type 5 (Soft blobs with clear cut edges passed easily), type 6 (Fluffy pieces with ragged edges, a mushy stool), and type 7 (watery, no solid pieces, entirely liquid).

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea, South Korea

IPD SHARING:
Plan to Share IPD: No